CLINICAL TRIAL: NCT04301765
Title: Improving Cancer-related Fatigue, Sexual Dysfunction and Quality of Life in Older Men With Cancer and Androgen Deficiency
Acronym: TEMEC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Principal Investigator, Jose Manuel Garcia, Principal Investigator, Seattle Institute for Biomedical and Clinical Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AG061558
Record Dates: First submitted 2020-03-03; First posted 2020-03-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hypogonadism, Male; Cancer; Fatigue
Keywords: testosterone; cancer related fatigue; active cancer; hypogonadism
MeSH Terms: conditions — Eunuchism; Neoplasms; Fatigue; Hypogonadism | interventions — Testosterone; Gels

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel group, trial of daily transdermal testosterone gel or placebo gel for 6-months
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- testosterone 1.62% gel (Experimental): Testosterone 1.62% gel will be applied daily by the participants (all participants will be trained in the application process and will be given printed instructions). The intervention will be for 6 months.
  Interventions: Drug: testosterone 1.62% gel
- placebo gel (Placebo Comparator): The placebo gel will be applied daily by the participants (all participants will be trained in the application process and will be given printed instructions). The intervention will be for 6 months.
  Interventions: Other: placebo gel

INTERVENTIONS:
Drug: testosterone 1.62% gel — The gel will be applied daily by the participants (all participants will be trained in the application process and will be given printed instructions). The intervention will be for 6 months
  Arms: testosterone 1.62% gel
Other: placebo gel — The gel will be applied daily by the participants (all participants will be trained in the application process and will be given printed instructions). The intervention will be for 6 months
  Arms: placebo gel

SUMMARY:
This is a large randomized, double-blind, placebo-controlled trial to determine the efficacy of testosterone replacement on cancer-related fatigue in older men with solid or hematologic (blood) cancer who report fatigue and have low testosterone levels.

DETAILED DESCRIPTION:
The overall objective is to conduct a double-blind, randomized, placebo-controlled, parallel group trial to determine the efficacy of 6 months of physiological testosterone replacement therapy in improving cancer related fatigue, sexual dysfunction, and body composition and muscle function in men 55 years and older with solid or hematologic (blood) cancers, who report fatigue and have testosterone deficiency. There will be 5 study visits: 1) Screening, 2) Baseline, 3) 2-Week Dose Adjustment Visit, 4) Three-month visit (Week 12), and 5) Six-month visit. Testosterone or placebo gels will be applied by eligible trial participants at home; participants will be trained on gel application procedures by research personnel.

ELIGIBILITY:
Inclusion Criteria:

* Men with active solid or hematologic (blood) cancers who have received or are receiving chemo- and/or radiation therapy. Patients who have no evidence of disease (NED) for 60 months or less, which means that they are <60 months from their last treatment (chemotherapy and/or radiation therapy) will be included.
* Age: 55 years and older
* Life expectancy of at least 6 months.
* Serum testosterone, measured by mass spectrometry (gold standard method), of <348 ng/dl and/or free testosterone <70 pg/ml. The lower limits of the normal range for total testosterone in healthy men is 348 ng/dL and the lower limits of free testosterone is <70 pg/ml in the Framingham Heart Study sample. As sex hormone binding globulin levels may be elevated in some men with cancer (resulting in elevation in total testosterone level), some of these symptomatic men may still be hypogonadal despite having total testosterone above this cut-off limit, but their free testosterone levels may still be below the lower limit of normal. Thus, men with free testosterone <70 pg/mL will be included.
* Fatigue. Fatigue was selected as it is a highly prevalent symptom in cancer patients. Fatigue will be defined as a score on FACIT-Fatigue subscale of <40, which best divides cancer patients from the general population with accuracy.
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Men with current or prior history of prostate, breast, testicular, or adrenal cancers.
* Use of anabolic agents (testosterone, DHEA, growth hormone) within the past 6 months
* Hematocrit >48%, serum creatinine >2.5 mg/dL
* PSA >4 ng/ml; nodule or induration on digital rectal exam
* Severe untreated sleep apnea
* Uncontrolled congestive heart failure
* Myocardial infarction, acute coronary syndrome, revascularization surgery, stroke or thromboembolism (of any etiology) within 6 months
* Known history of thrombophilia due to a genetic mutation (e.g. Factor V Leiden)
* Previous stroke with residual cognitive or functional deficits
* Inability to provide informed consent; MMSE score <24
* Poorly controlled diabetes as defined by hemoglobin A1c >10.0%
* Body mass index (BMI) >40 kg/m2
* Bipolar disorder or schizophrenia

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-01-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue change | 6 months
  Primary outcome is change in fatigue score. Fatigue will be assessed by the Functional Assessment of Chronic Illness Therapy fatigue scale (FACIT-Fatigue)- The FACIT-Fatigue has been widely used in studies related to cancer-related fatigue and is able to detect clinically meaningful differences in fatigue scores in response to treatment. Population norms for the FACIT are also available, facilitating the interpretation of fatigue levels in patient populations. This instrument has been well-validated, is responsive to treatment and more sensitive to change in fatigue than other instruments. Score range: 0-52, the higher the score the better quality of life.

SECONDARY OUTCOMES:
Change in Sexual Activity Score | 6 months
  Secondary outcome is change in sexual activity score, assessed by the Harbor-UCLA 7-day Sexual Function Questionnaire.

OTHER OUTCOMES:
Change in Other Measures of Sexual Function | 6 months
  Erectile function will be assessed by International Index of Erective Function (IIEF).
Change in Mood and Well-being | 6 months
  Mood and well-being will be assessed by Positive and Negative Affect Scale (PANAS), which includes 10 questions each for Positive Affect and Negative Affect. Many behavioral scientists consider affectivity as the cleanest window on an individual's wellbeing. The most sensitive indicator of impaired wellbeing has been shown to be affective dysregulation, which is reflected in affectivity balance. The latter incorporates negative affects (e.g., anxiety, depression) as well as positive affects (e.g., joy).
Body Composition Changes | 6 months
  Body composition changes will be assessed by measuring lean body mass and fat mass by dual energy X-ray absorptiometry (DEXA).
Muscle Strength Changes | 6 months
  Muscle strength will be assessed by measuring maximal voluntary strength in the leg press exercise by the 1-RM method.
Physical Function Changes | 6 months
  Physical function will be evaluated using the 6-minute walk test and will also be evaluated by measuring power in the lower extremities by conducting the leg press exercise.
Objective Measures of Habitual Physical Activity Changes | 6 months
  To determine changes in daily physical activity, validated actigraphy will be used.
Caregiver Burden Changes | 6 months
  The Brief Assessment Scale for Caregivers (BASC) will be used to determine caregiver burden.
Work Productivity | 6 months
  Loss of productivity will be evaluated using the Work Productivity and Impairment (WPAI) scale.
Sleep Quality Changes | 6 months
  Sleep quality will be assessed using the validated Pittsburgh Sleep Quality Index (PSQI) scale and by using actigraphy.
Qualitative Survey | 6 months
  Qualitative interviews will be performed by a study co-investigator which will assess lived experiences of participants at baseline and at 24 weeks by conducting semi-structured, qualitative phone interviews with a randomly selected sample of 30 men in the testosterone arm and 30 men in the placebo arm (equally divided across the 3 sites).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No